CLINICAL TRIAL: NCT05851768
Title: Analgesic Efficacy of Adding Dexmedetomidine VS Magnesium Sulphate as Adjuvants With Bupivacaine in Ultrasound-guided Erector Spinae Plane Block for Post Thoracotomy Pain
Brief Title: Efficacy of Dexmedetomidine VS Magnesium Sulphate With Bupivacaine in Erector Spinae Block for Thoracotomy Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Walaa Youssef Elsabeeny, Assistant professor of Anesthesia and Pain management, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N-80-2022/NSC
Record Dates: First submitted 2023-05-01; First posted 2023-05-10 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia | interventions — Bupivacaine; Magnesium; Dexmedetomidine

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Masking Description: Double blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Erector spinae plane block with 0.25% bupivacaine (Active Comparator): Patients will receive ultrasound guided ESPB with 0.25% bupivacaine
  Interventions: Drug: Bupivacaine
- Erector spinae plane block with 0.25% bupivacaine and Magnesium (Experimental): Patients will receive ultrasound guided ESPB with 0.25% bupivacaine and magnesium
  Interventions: Drug: Bupivacaine + Magnesium
- Erector spinae plane block with 0.25% bupivacaine and Dexmedetomidine (Experimental): Patients will receive ultrasound guided ESPB with 0.25% bupivacaine and dexmedetomidine
  Interventions: Drug: Bupivacaine + Dexmedetomidine

INTERVENTIONS:
Drug: Bupivacaine — Bupivacaine 0.25%
  Arms: Erector spinae plane block with 0.25% bupivacaine
Drug: Bupivacaine + Magnesium — Bupivacaine 0.25% + Magnesium
  Arms: Erector spinae plane block with 0.25% bupivacaine and Magnesium
Drug: Bupivacaine + Dexmedetomidine — Bupivacaine 0.25% + Dexmedetomidine
  Arms: Erector spinae plane block with 0.25% bupivacaine and Dexmedetomidine

SUMMARY:
Postoperative pain management is considered an integral part of perioperative care in patients undergoing thoracotomy. In order to reduce these complications, multiple regional techniques have been developed for thoracotomy including Intercostal nerve block, Erectospinae plane block and serratus block. Multiple adjuvants have been used in regional analgesia including adrenaline,clonidine,magnesium sulphate,dexmedatomidine and opoids.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 65 years.
* Male and female sexes.
* ASA I-II.,III
* Cancer patients undergoing thoracotomy incisions
* Body mass index (BMI) from 18.5 to 30 kg/m2

Exclusion Criteria:

* Patient refusal
* Known allergy to any of the used drugs
* Low platelet count, any coagulation defect

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-03-25 (Estimated); Study Completion 2024-04-27 (Estimated)

PRIMARY OUTCOMES:
Total postoperative morphine consumption | First 24 hours postoperatively
  Total dose of morphine needed postoperatively in the first 24 h

SECONDARY OUTCOMES:
Time to first postoperative rescue analgesia. | First 24 hours postoperatively
  Time to first postoperative rescue analgesia.

CONTACTS AND LOCATIONS:
Overall Officials: Walaa Y Elsabeeny, MD, Principal Investigator — Assistant professor of Anesthesia and Pain Management, National Cancer Institute, Cairo University; Ahmed A Mohamed, MD, Study Director — Professor of Anesthesia,Surgical intensive care and Pain management,Faculty of medicine
Locations (1):
- Walaa Y Elsabeeny, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Information is available upon reasonable request through contacting the corresponding investigator